CLINICAL TRIAL: NCT02108730
Title: Towards Individualized Surgery in Non-focal Congenital Hyperinsulinism
Acronym: non-focal CHI
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Prof. Winfried Barthlen, Professor of Pediatric surgery, University Medicine Greifswald
Other Study IDs: 123456
Record Dates: First submitted 2014-03-28; First posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Non-focal Congenital Hyperinsulinism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- non-focal congenital hyperinsulinism: 13 children and one adult with non-focal congenital hyperinsulinism
  Interventions: Procedure: restrictive pancreatic resection

INTERVENTIONS:
Procedure: restrictive pancreatic resection — Restrictive, spleen-preserving resection of the pancreatic tail by laparoscopy

SUMMARY:
Observational study in patients with non-focal congenital hyperinsulinism showing that restrictive surgery may improve the metabolic situation

DETAILED DESCRIPTION:
In non-focal congenital hyperinsulinism (CHI) the current doctrine warrants subtotal pancreatic resection in all children who do not respond to medication. However, the rate of diabetes after these extensive resections is very high. In this study investigators show that a less aggressive approach may suffice to wean many children from all medication or to get them manageable medically.

ELIGIBILITY:
Inclusion Criteria:

* patients with non-focal congenital hyperinsulinism

Exclusion Criteria:

* patients with focal congenital hyperinsulinism

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 13 children and one adult (30 years)
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
necessity of medication after restrictive surgery in congenital hyperinsulinism | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Barthlen, Professor of Pediatric Surgery, Principal Investigator — University Medicine Greifswald
Locations (1):
- Pediatric Surgery, Greifswald, Germany

REFERENCES:
- See also: homepage of Pediatric Surgery in Greifswald, Germany — http://www.medizin.uni-greifswald.de/ki_chir/index.php?id=14&L=1